CLINICAL TRIAL: NCT06465667
Title: Improving Engagement With a Process Measure Dashboard Through Precision Feedback
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Kristian Stensland, Assistant Professor of Urology, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: HUM00248876
Record Dates: First submitted 2024-06-13; First posted 2024-06-20 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Behavior
Keywords: Ureteral stent omission; Ureteral stent placement; Behavior change; Dashboard; Precision feedback
MeSH Terms: conditions — Behavior | interventions — Dashboard Systems

STUDY DESIGN:
Intervention Model Description: This is be a stepped wedge randomized controlled trial of precision feedback. One hundred urologists will be randomized into four groups, stratified by case volume. The trial will consist of four steps of three months each, at the beginning of which one group will cross over from control to intervention arm. This is preceded by a three-month pre-rollout period, comprising a total study length of 15 months. The duration of the trial was chosen based on a desire to deliver "rapid" results to inform the scale-up of the intervention, and to mirror the period of time over which a typical dashboard project may be conceived, designed, and delivered. Case volume may predict dashboard engagement, stenting practices, and privileged awareness of ongoing study efforts, and is therefore suitable for stratification.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 dashboard (3 months) then dashboard with Precision feedback (12 months) (Experimental): Months 0-3 dashboard only, months 3-15 months dashboard with Precision feedback.
  Interventions: Behavioral: Dashboard; Behavioral: Precision Feedback Push
- Group 2 dashboard (6 months) then dashboard with Precision feedback (6 months) (Experimental): Months 0-6 dashboard only, months 6-15 months dashboard with Precision feedback.
  Interventions: Behavioral: Dashboard; Behavioral: Precision Feedback Push
- Group 3 dashboard (9 months) then dashboard with Precision feedback (6 months) (Experimental): Months 0-9 dashboard only, months 9-15 months dashboard with Precision feedback.
  Interventions: Behavioral: Dashboard; Behavioral: Precision Feedback Push
- Group 4 dashboard (12 months) then dashboard with Precision feedback (3 months) (Experimental): Months 0-12 dashboard only, months 12-15 months dashboard with Precision feedback.
  Interventions: Behavioral: Dashboard; Behavioral: Precision Feedback Push

INTERVENTIONS:
Behavioral: Dashboard — The Dashboard intervention, representing current standard of care, will consist of a standard e-mail message with a link to the dashboard and text explanation. No performance data will be included in the e-mail, and links will not be monitored for clickthrough with repeat e-mail.
Behavioral: Precision Feedback Push — The experimental intervention, precision feedback e-mail messaging, will consist of an e-mail with a link to the dashboard along with tailored information about a participant's performance in the quality process measure of interest. For example, e-mail subject lines may read "You have room for improvement in stent omission," accompanied by a visual display in the body of the e-mail showing a participant's performance relative to a top performing peer. The behavior change intervention delivery component will also involve modifications to existing procedures. Namely, performance feedback will be reported directly in the e-mail as either plain text, or an embedded or attached image with graphed data.

SUMMARY:
The study seeks to assess the impact of e-mailing specific, targeted, practice-pattern based information ("precision feedback") on provider engagement with a dashboard for a quality process measure (showing stent omission after pre-stented ureteroscopy), compared with generic information ("one size fits most" feedback).

DETAILED DESCRIPTION:
The Michigan Urological Surgery Improvement Collaborative (MUSIC) is a state-wide, physician-led quality improvement collaborative comprised of over 40 urology practices representing varied practice sites within Michigan and nationally, designed to evaluate and improve the quality of urologic care.

A recently identified area for quality improvement within MUSIC is avoidance of placing ureteral stents following uncomplicated ureteroscopy and lithotripsy for kidney stones. Such unnecessary stents do not measurably increase post-operative safety, but rather have been shown to contribute to unnecessary emergency department visits. This process measure (stent omission after uncomplicated ureteroscopy) is the subject matter for the dashboard and will serve as the focus of precision feedback.

The study team hypothesizes that a behavior change intervention bundle consisting of "precision feedback" along with communication strategies to simplify access to feedback will increase dashboard engagement (measured via click-through rate and dashboard logins) compared with standard "one size fits most" e-mail messages. Knowledge gained from this study will inform the development of other precision feedback programs within our urology quality improvement collaborative (MUSIC), and provide a framework for rapid, pragmatic trials for small to mid-sized collaborative quality initiatives nationally.

ELIGIBILITY:
Inclusion Criteria:

-Urologists participating in MUSIC that were in the top one hundred individuals in annual case volume from 2023 for "pre-stented ureteroscopy", the case for which the dashboard contents are most relevant.

Exclusion Criteria:

- Urologists that are not in the top one hundred individuals in annual "pre-stented ureteroscopy" case volume, urologists in the study team, or that opt out from the study at the individual or site level.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-07-17 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Clickthrough rate to the online dashboard | Every 3 months up to 15 months
  Clickthrough is defined as a link ever being clicked in the three months following e-mail send date, at which point in time a new e-mail will be sent. Clickthrough rate will be calculated as the number of clickthroughs divided by number of links sent (i.e., opportunities for clickthrough).

SECONDARY OUTCOMES:
Total number of dashboard visits | 15 months
  Dashboard visits captured by Google Analytics.
Cumulative time (minutes) spent on the dashboard | 15 months
  Time spent will be captured by Google Analytics.
Urologist opt-out rate | 15 months
Helpful/not helpful rate | 15 months
  There will be one question if the intervention was helpful or not.
Stent rate for pre-stented ureteroscopy | 15 months
E-mail open rate | Every 3 months up to 15 months
  E-mail open rate will be measured as number of e-mail opens divided by number of e-mails sent.

CONTACTS AND LOCATIONS:
Overall Officials: Kristian Stensland, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lewicki P, Clark S, Shoemaker E, Wang B, Ross J, Daignault-Newton S, Carlozzi N, Martin-Schwarze A, Meurer W, Sales A, Ghani K, Dauw C, Stensland K. Rationale and protocol for a prospective clinical trial enrollment improvement hybrid study within a trial. Contemp Clin Trials Commun. 2025 Sep 20;48:101548. doi: 10.1016/j.conctc.2025.101548. eCollection 2025 Dec. PMID 41050879
- [Derived] Lewicki P, Salka B, Daignault-Newton S, Ross J, Krumm A, Ghani KR, Dauw C, Landis-Lewis Z, Stensland KD; Michigan Urological Surgery Improvement Collaborative. Rapid cycle, randomised testing of precision feedback to improve engagement with a process measure dashboard amongst urologists: study protocol for a hybrid trial. BMJ Open. 2025 May 6;15(5):e092742. doi: 10.1136/bmjopen-2024-092742. PMID 40335130